CLINICAL TRIAL: NCT06332495
Title: Research Project on the Risk of Discomfort, Pain and Alteration of Skin Condition in Bedpan Use by Patients and Caregivers
Brief Title: Research Project on the Risk of Discomfort, Pain, Alteration of Skin Condition in Bedpan Use by Patients and Caregivers
Acronym: RIDAECUBA
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC23_0573; 2024-A00025-42 (Other: ANSM (IDRCB))
Record Dates: First submitted 2024-03-13; First posted 2024-03-27 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Nurse-Patient Relations
Keywords: Bedpan; Discomfort; Alteration of Skin; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Assessment of pain during pelvic positioning: 48-hour follow-up of patients included in the study, with data collected on two pelvis fittings per 24 hours of follow-up (one fitting = one installation and one removal).
  Interventions: Other: Questioning the patient during hygiene care

INTERVENTIONS:
Other: Questioning the patient during hygiene care — The study examines how patients and caregivers feel when using the bedpan. Over the course of a day, collecting all this information would take just under 7 minutes. Over the duration of patient participation (2 days), we estimate that it would take a total of 15 minutes per patient to collect this information. The objectives are focused on pain and discomfort, and on the alteration of the (patient's) skin condition through objective observation of redness or stage I pressure sores by the caregiver.

SUMMARY:
The hypothesis is that the current bedpan is not adapted to the diversity of patients encountered. It is necessary to collect the opinions of patients themselves on the current pool in different departments in order to validate our hypothesis.

The objective is to evaluate pain in patients with reduced or very reduced mobility caused by the bedpan currently used in current practice through an observational study.

DETAILED DESCRIPTION:
Patients with reduced or severely reduced mobility, over 18 years of age, bedridden and requiring the use of a bedpan, estimated hospitalization equal to or greater than 2 days on the ward.

ELIGIBILITY:
Inclusion Criteria:

* Patient of legal age (age ≥ 18 years).
* Patient with reduced and very reduced mobility, bedridden requiring the use of a bedpan.
* Estimated length of hospital stay on the ward ≥ 2 days.
* Patient affiliated to a social security system.
* Patient able to understand the protocol.
* Patient having given oral non-opposition to participate.
* Patient who has received the study information note.
* Patient who had never participated in this study.

Exclusion Criteria:

* Patients with cognitive impairment preventing objective pain assessment or with neurological pathologies.
* Patients under guardianship, curatorship or safeguard of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with reduced or severely reduced mobility, over 18 years of age, bedridden and requiring the use of a bedpan, estimated hospitalization equal to or greater than 2 days.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-08-03 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-03 (Estimated)

PRIMARY OUTCOMES:
Assessment of pain in a patient with reduced or very reduced mobility when using a bedpan. | Four assessments in 48 hours
  Pain will be assessed using a numerical pain scale (EN). The caregiver will ask the patient to rate his or her pain between 0 (no pain) and 10 (the most intense pain imaginable).

SECONDARY OUTCOMES:
Assess the proportion of patients with a MCID of the pain felt by the patient in pre-installation > 1.3 | 48 hours
Assess the maximum pain felt by the patient pre/post and per/post use of the bedpan. | 48 hours
  Pain will be assessed using a numerical pain scale (EN). The caregiver will ask the patient to rate his or her pain between 0 (no pain) and 10 (the most intense pain imaginable).
Assess patient discomfort on the bedpan | 48 hours
  discomfort will be defined by the addition of a cushion, rolled towel, treatment oil or the need for the bedpan to be repositioned
Assess alteration of skin condition at the seat of the patient using the bedpan | 48 hours
  Appearance of stage I redness or pressure sores (redness that does not disappear) on the patient's seat, after using the bedpan
Assess the caregiver's pain when handling the bedpan, placing the bedpan in position and removing the bedpan. | 48 hours
  Pain will be assessed using a numerical pain scale (EN). The caregiver will rate his or her pain between 0 (no pain) and 10 (the most intense pain imaginable).
Assess the risk factors associated with the onset of pain when placing a bedpan. | 48 hours
Assess the difficulty of positioning and removing the bedpan. | 48 hours
  Painfulness of placing and removing the bedpan, assessed by the caregiver using a Likert scale between 1 (easy) and 5 (impossible alone)
Assess bedpan stability during use | 48 hours
  Stability will be evaluated by the tilting, or not, of the bedpan during use by the patient.
Evaluate the effect of time spent on the bedpan on: pain, skin alteration and discomfort | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pia SECHER, Principal Investigator — Nantes University Hospital
Locations (5):
- France (5):
  - Nantes University Hospital, Nantes, Loire Atlantique
  - CHU Cholet, Cholet
  - CHU Laval, Laval
  - CH Le Mans, Le Mans
  - CHU Orleans, Orléans

IPD SHARING:
Plan to Share IPD: No